CLINICAL TRIAL: NCT01227694
Title: Articular Cartilage Regeneration in Gonarthrosis Grade II and III by Articular Infiltration of Xcel-m-condro-alpha.
Brief Title: Adult Stem Cell Therapy for Repairing Articular Cartilage in Gonarthrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Banc de Sang i Teixits (Other)
Collaborators: Centro Medico Teknon (Other); Institut de Terapia Regenerativa Tissular (Other); Cetir Sant Jordi, S.a.. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XCEL-M-09-01
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Osteoarthritis, Knee; Knee Injuries; Joint Diseases; Rheumatic Diseases; Cartilage Diseases
Keywords: Cell therapy; Regenerative therapy; Advance therapy; Bone marrow; Mesenchymal stem cell; Autologous; Interventional clinical trial; Osteoarthrosis; Osteoarthritis; Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Knee Injuries; Joint Diseases; Rheumatic Diseases; Cartilage Diseases; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous MSC knee implantation (Experimental): Isolation and "Ex-Vivo" expansion of Mesenchymal stem cells (MSC) obtained from each patient's bone marrow under GMP conditions at Xcelia-División de Terapias Avanzadas del Banc de Sang I Teixits. After 21 days, approximately 40 millions of autologous MSC will be implanted in the knee by articular injection.
  Interventions: Other: Autologous MSC knee implantation

INTERVENTIONS:
Other: Autologous MSC knee implantation — Isolation and "Ex-Vivo" expansion of Mesenchymal stem cells (MSC) obtained from each patient's bone marrow under GMP conditions at Xcelia-División de Terapias avanzadas del Banc de Sang I Teixits. After 21 days, approximately 40 millions of autologous MSC will be implanted in the knee by articular injection.
  Other Names: Xcel-m-condro-alpha

SUMMARY:
This is a prospective, open-label, single-dose, single-arm phase I-II study in which 15 patients diagnosed with gonarthrosis grade II-III (Kellgren and Lawrence) will enter the study with the primary objective of assessing the feasibility and safety of the knee articular infiltration of autologous bone marrow mesenchymal stem cells (MSC). Secondary objectives are to assess the efficacy by imaging procedures and clinical questionnaires.

MSC obtained from each patient's bone marrow will be isolated and expanded "Ex-Vivo" under GMP conditions at Xcelia-División de Terapias avanzadas del Banc de Sang I Teixits. After 21 days, patients will be implanted a single-dose of approximately 40 millions of autologous MSC in the knee by articular injection, and followed up for 12 month. Articular cartilage changes will be determined by T2-weighted MRI (Cartigram) at 6 and 12 month. Clinical assessment will measure the pain by the visual analogue scale (VAS), the self-reported functional status by Heath Assessment Questionnaire (HAQ), and the quality of life by Short Form 36 questionnaire (SF-36) at 3, 6 and 12 month.

The working hypothesis proposes that the expected regenerative articular cartilage effect of the MSC will be produced to a measurable degree by imaging procedures and clinical questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Gonarthrosis grade II-III of Kellgren and Lawrence assessed by two observers
2. Chronic knee pain with mechanical characteristics
3. Absence of local or systemic septic process
4. Haematological and biochemical laboratory tests without significant alterations that contraindicate treatment.
5. Informed Consent form signed by the patient
6. The patient is able to understand the nature of the study

Exclusion Criteria:

1. Patients < 18 years or legally dependent
2. Patients >65 years
3. Previous surgery of the knee
4. Intraarticular treatment in the past 6 month
5. Knee ligament or meniscus rupture observed by MRI
6. Any sign of infection
7. Positive serology for HIV-1 or HIV-2, Hepatitis B (HBsAg), Hepatitis C (Anti-HCV-Ab) and syphilis.
8. Congenital or acquired malformation resulting in significant deformity of the knee and leading to problems in application or evaluation of results.
9. Overweight expressed as body mass index (BMI) greater than 30.5 (obesity grade II). BMI estimated as mass (kg) / corporal surface (m2).
10. Pregnant women or intend to become pregnant or breast-feeding
11. Neoplasia
12. Immunosuppressive states
13. Participation in another clinical trial or treatment with a different investigational product within 30 days prior to inclusion in the study.
14. Other pathologic conditions or circumstances that difficult participation in the study according to medical criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of autologous bone marrow mesenchymal stem cells (MSC) knee articular infiltration. | 12 months
  Feasibility will be assessed by checking the cascade of procedures (from bone marrow extraction to MSC implantation) and confirming the global process is viable.
Safety of autologous bone marrow mesenchymal stem cells (MSC) knee articular infiltration. | 12 months
  Safety will be assessed by collecting adverse events throughout the experimental phase, including the follow-up at 12 months.

SECONDARY OUTCOMES:
Efficacy by imaging procedures. | 6 months
  Articular cartilage changes will be determined by T2-weighted MRI (Cartigram).
Efficacy by imaging procedures. | 12 month
  Articular cartilage changes will be determined by T2-weighted MRI (Cartigram).
Clinical outcomes. | 3 month
  Clinical assessment will measure the pain by the visual analogue scale (VAS), the self-reported functional status by Heath Assessment Questionnaire (HAQ), and the quality of life by Short Form 36 questionnaire (SF-36).
Clinical outcomes. | 6 months
  Clinical assessment will measure the pain by the visual analogue scale (VAS), the self-reported functional status by Heath Assessment Questionnaire (HAQ), and the quality of life by Short Form 36 questionnaire (SF-36).
Clinical outcomes. | 12 months
  Clinical assessment will measure the pain by the visual analogue scale (VAS), the self-reported functional status by Heath Assessment Questionnaire (HAQ), and the quality of life by Short Form 36 questionnaire (SF-36).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Soler, MD, Principal Investigator — Institut de Teràpia Regenerativa Tissular (ITRT)
Locations (1):
- Centro Medico Teknon-ITRT, Barcelona, Spain

REFERENCES:
- [Derived] Vives J, Oliver-Vila I, Pla A. Quality compliance in the shift from cell transplantation to cell therapy in non-pharma environments. Cytotherapy. 2015 Aug;17(8):1009-14. doi: 10.1016/j.jcyt.2015.02.002. Epub 2015 Mar 10. PMID 25769789
- See also: Institut de Terapia Regenerativa Tissular (ITRT), Barcelona, Spain — http://www.itrt.es
- See also: Banc de Sang i Teixits — http://www.bancsang.net